CLINICAL TRIAL: NCT02751840
Title: Effects of Caffeine and Coffee on Resting Metabolic Rate, Comparing Normal Weight Men to Obese Men
Acronym: RMR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Tel Hai College RMR-011
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Asymptomatic Conditions
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Caffeine; Coffee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caffeine (Experimental): Caffeine capsule (200 mg) is taken prior to RMR measurement
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Placebo; Other: Coffee; Other: Decaffeinated
- Placebo (Placebo Comparator): Placebo (starch) capsule is taken prior to RMR measurement
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Placebo; Other: Coffee; Other: Decaffeinated
- Coffee (Experimental): Black coffee (9 grams) is consumed prior to RMR measurement
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Placebo; Other: Coffee; Other: Decaffeinated
- Decaffeinated (Placebo Comparator): Decaffeinated Black coffee (9 grams) is consumed prior to RMR measurement
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — 200 mg of caffeine capsule before RMR measurement
Dietary Supplement: Placebo — Placebo capsule (starch) before RMR measurement
Other: Coffee — 9 grams of black coffee in boiling water consumed before RMR measurement
  Arms: Caffeine; Coffee; Placebo
Other: Decaffeinated — 9 grams of decaffeinated black coffee in boiling water consumed before RMR measurement
  Arms: Caffeine; Coffee; Placebo

SUMMARY:
Background. The prevalence of obesity has increased in the last two decades. To maintain body weight energy expenditure (EE) should be equal to energy intake (EI). A low EE predisposes individuals to weight gain and to obesity that can also results from low resting metabolic rate (RMR). Caffeine (Caf) is an active food ingredient and is widely consumed globally, and has an important impact on energy balance. Caf reduces appetite (EI) and increases EE, thus, Caf has a potential role in body weight reduction. Caf causes higher total daily energy expenditure (TDEE) in normal weight (NW) people compared to obese (OW). Moreover Caf is linked to decreased fat oxidation in OW. There are differences between OW and NW in Caf pharmacokinetics, but no differences reported between NW and OW females in its effects on RMR. There is a gender difference in the influence of Caf on metabolism. The investigators are aware of no previous studies which compared the effect of Caf on the RMR of NW and OW men.

Objectives. 1) To compare the effect of Caf and coffee on resting metabolic rate (RMR) values in healthy normal-weight (NW) men and overweight (OW) men. 2) To develop Caf intake frequency questionnaire (in Hebrew)

Hypothesis. RMR values will be higher and respiratory exchange ratio (RER) values will be lower in NW compared to the values measured in OW men.

Methods. 33 men (16 NW and 17 OW) were reported to the laboratory on 4 separate occasions (placebo, Caf tablets, coffee and decaffeinated coffee). During the lab sessions they were undergo complete anthropometric measurements and RMR measured (one of the study conditions) using indirect calorimetry. Additionally, respiratory exchange ratio (RER) which is calculated as the ratio between CO2 production (VCO2) and O2 consumption (VO2) (VCO2/VO2), blood pressure and heart rate (HR) response recorded.

The importance of this study is that the results will contribute to the scientific basis of weight control and health interventions programs (diet and physical activity) in overweight men.

DETAILED DESCRIPTION:
Methods. 16 NW and 17 OW men were reported to the laboratory on 4 separate occasions (placebo, Caf tablets, coffee and decaffeinated coffee) each separated by 2-7 days. Before the first meeting they refill caffeine, physical activity and medical questionnaires. The investigators recruited only men who were healthy non-smokers with no comorbidities and the daily caffeine consumption was under 400 mg. Before each meeting participants had to comply guidelines outlined included fasting for 8 hours, avoiding intense physical activity 14 hours and moderate exercise 2 hours before measurements. The meetings conducted in the morning when the first session included anthropometric measurements (weight, height and waist circumference) and body composition measurements using Bioelectrical Impedance Analysis (BIA) and a digital caliper. Each session began with a measuring resting blood pressure and heart rate (Polar telemetric systems), after that participants were given randomly placebo or Caf tablets or coffee or decaffeinated coffee, waiting half an hour and then measuring the RMR and respiratory exchange ratio (RER), for half an hour using indirect calorimetry (canopy system). Then again measured blood pressure and heart rate at rest.

The sample size was calculated for 16 participant in each group, according to an expected change of 3% at RMR values between the groups with the power of 80% and significance of 0.05 . standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

33 Healthy men at the age between 20-50 years. 16 normal weight men and 17 obese men.

Exclusion Criteria:

1. Hypertension (above 140/90 mmHg)
2. Taking medications for hypertension
3. Heart, liver or kidney problems, diabetes, respiratory problems, hypo/hyper thyroidism.
4. Smoking
5. Men who consume caffeine above 400 mg/day
6. Taking medications or dietary supplements that can affect energy expenditure
7. Elite athletes (competitive sport)
8. Night Eating

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Measurement of resting metabolic expenditure using indirect calorimetry (open flow canopy system) | Within two weeks (4 sessions, each 30 minutes)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acheson KJ, Zahorska-Markiewicz B, Pittet P, Anantharaman K, Jequier E. Caffeine and coffee: their influence on metabolic rate and substrate utilization in normal weight and obese individuals. Am J Clin Nutr. 1980 May;33(5):989-97. doi: 10.1093/ajcn/33.5.989. PMID 7369170
- [Background] Adan A, Prat G, Fabbri M, Sanchez-Turet M. Early effects of caffeinated and decaffeinated coffee on subjective state and gender differences. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Oct 1;32(7):1698-703. doi: 10.1016/j.pnpbp.2008.07.005. Epub 2008 Jul 15. PMID 18675877
- [Background] Bracco D, Ferrarra JM, Arnaud MJ, Jequier E, Schutz Y. Effects of caffeine on energy metabolism, heart rate, and methylxanthine metabolism in lean and obese women. Am J Physiol. 1995 Oct;269(4 Pt 1):E671-8. doi: 10.1152/ajpendo.1995.269.4.E671. PMID 7485480
- [Background] Jeukendrup AE, Randell R. Fat burners: nutrition supplements that increase fat metabolism. Obes Rev. 2011 Oct;12(10):841-51. doi: 10.1111/j.1467-789X.2011.00908.x. PMID 21951331
- [Background] Temple JL, Ziegler AM. Gender Differences in Subjective and Physiological Responses to Caffeine and the Role of Steroid Hormones. J Caffeine Res. 2011 Mar;1(1):41-48. doi: 10.1089/jcr.2011.0005. PMID 24761262
- [Background] Pohanka M. The perspective of caffeine and caffeine derived compounds in therapy. Bratisl Lek Listy. 2015;116(9):520-30. doi: 10.4149/bll_2015_106. PMID 26435014